CLINICAL TRIAL: NCT02038413
Title: In Silico Clinical Trial, Comparing State of the Art Photon Modalities With Proton and 12C-ion Therapy for Stage I NSCLC: A Multicentric ROCOCO Planning Study Based on a Reference Dataset of Patients
Brief Title: State of the Art Photon Therapy Versus Particle Therapy for Small Lung Tumors; a Planning Study Based on a Reference Dataset of Patients
Acronym: Lung stage I
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: ROCOCO Lung stage I
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; cT1/cT2aN0M0; Stereotactic lung treatment; MAASTRO; age >18 years
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC stage I: Consecutive patients were identified from October 2009 onwards in MAASTRO clinic, Maastricht. All patients received respiratory gated CT (4DCT) scans. All were patients referred for primary radiotherapy or chemo radiation.

SUMMARY:
Compared to conventional radiotherapy with photons (CRT), particle therapy (PT) has the potential to inflict maximum damage on tumors with minimum collateral damage to neighboring healthy tissue. Given that the cost of particle therapy (PT) is considerably higher than that of conventional radiotherapy (RT) with photons, it is necessary to establish whether these higher costs are worthwhile in light of the expected advantages. Thus, clear evidence of the situations in which PT outperforms conventional photon treatment is needed.

In a previous ROCOCO study (lung stage I-IIIB) an inhomogeneous group of patients with regard to tumor stage and size was included1. Conformal radiotherapy and Intensity Modulated Radiotherapy were used in the comparison. In this study patients with smaller tumors are included (stage I). A stereotactic treatment schedule and more advanced treatment techniques, such as CyberKnife, RapidArc, IMRT and Tomotherapy, are eligible for these kind of lesions. As a result the comparison as demonstrated in our previous study maybe invalid. We propose to investigate to what extend proton and 12C-ion therapy decrease the amount of irradiated normal tissue compared to state of the art photon modalities in stage I lung cancer patients.

DETAILED DESCRIPTION:
For this in silico planning study all treatment plans will be performed in centers that are already operating and have experience in treatment planning. IMRT treatment plans will be calculated in Eindhoven (NL), Tomotherapy plans in Deventer (NL), Cyberknife plans in Liege (BE) and RapidArc treatment plans in Hasselt (BE). Proton treatment plans will be performed at the University of Pennsylvania (USA) and the C-ion treatment plans at the University of Marburg (GE).

A dataset with state-of-the-art image data is available. 25 patients will be included according to a-priori defined selection criteria. Each patient will function as his or her own control. For this reason, the number of patients per tumor group can be limited to 25 patients per tumor group (power = 80%, alpha = 5%).

The datasets will be stored on a secure website hosted by MAASTRO. High quality CT-images will be used for radiotherapy treatment planning. Secondary image information such as FDG-PET and MRI will be used for GTV delineation. GTV and all relevant OARs will be delineated in MAASTRO (NL). The GTV to PTV margin will be determined by the individual institutes according to the treatment technique and treatment modality.

Photons will be planned with state of the art treatment techniques. Protons will be planned using active beam delivery with Intensity Modulated proton therapy (IMPT)and carbon-ions with a pencil beam delivery treatment planning technique with gantry. Each participating center will use its own treatment planning system according to standard practice at that center. The same tumor dose, overall treatment time (OTT) and an equal number of fractions will be used for all treatment modalities.

Photon, proton and C-ion treatments will be compared based on dosimetric parameters on normal tissues. DVH's will be calculated for the OARs. In addition, the NTCP for a fixed tumor dose will be determined. Cobalt Gy equivalent doses will be used when reporting the proton and carbon-ion dose. In the case of protons, a constant RBE value of 1.1 will be used for both the tumor and the normal tissues. The RBE of carbon-ions will be calculated based on the models used by the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* referred for primary radiotherapy or chemo radiation
* NSCLC stage I
* received respiratory gated CT (4DCT) scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 25 NSCLC patients; stages I (cT1/cT2aN0M0). Consecutive patients were identified from October 2009 onwards in MAASTRO clinic, Maastricht. All patients received respiratory gated CT (4DCT) scans. All were patients referred for primary radiotherapy or chemo radiation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Radiation exposure for organs at risk (OAR) in a stereotactic lung radiotherapy treatment. | 1 year
  A wide range of organs is included, to be able to document doses to organs that are further away from the target volume, and also to quantify low doses to organs.
  Included OAR's are; left lung, right lung, (part of the) ribs if less then 2 cm from the CTV, for non-apical tumors: liver, spinal canal resembling the spinal cord, esophagus (full length), trachea, and main bronchi up to the first bifurcation, skin (with a thickness of standardized 4 mm), thyroid area, heart, mediastinal great vessels (aorta, vena cava, main lung arteries, ...), portacath, pacemaker (or any other implanted device to be avoided), brachial plexus and stomach.

SECONDARY OUTCOMES:
The risk of side effects in the irradiated normal tissue | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands; Esther Troost, PhD, Study Director — Maastro Clinic, The Netherlands; Erik Roelofs, Study Director — Maastro Clinic, The Netherlands; Esther Bloemen, Study Director — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands